CLINICAL TRIAL: NCT02051569
Title: Everyday Social Behavior and Mood in Individuals With a Family History of Depression. Investigating the Role of Serotonin
Brief Title: Serotonin and Everyday Social Interaction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Marije aan het Rot, Assistant Professor, University of Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL451-09-013 / 2
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Social Behaviour
MeSH Terms: conditions — Social Behavior | interventions — Tryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tryptophan first (Experimental): Tryptophan is given for the first 14 days, 6 times 500mg per day. Placebo is given 6 times per day for the second 14 days.
  Interventions: Dietary Supplement: Tryptophan
- Tryptophan second (Experimental): Placebo is given 6 times per day for the first 14 days. Tryptophan is given for the second 14 days, 6 times 500mg per day.
  Interventions: Dietary Supplement: Tryptophan

INTERVENTIONS:
Dietary Supplement: Tryptophan — Tryptophan and placebo are given in a crossover design, based on randomisation.

SUMMARY:
Rationale: Poor social functioning may contribute to major depressive disorder (MDD). Poor serotonin function may also contribute to MDD. Recent research suggests that serotonin plays a role in regulating human social behaviour. Therefore it would be intriguing to investigate the role of serotonin in regulating the quality of everyday social interactions in a population at risk for MDD. Human social behaviour can be reliably assessed in everyday life using Ecological Momentary Assessment (EMA).

Objective: This study aims to investigate how an experimental increase in serotonin influences social functioning in healthy adults with a first-degree family member diagnosed with MDD. The primary goal is to investigate the role of serotonin in regulating everyday social behaviour, measured using EMA. This will be done using oral supplementation with tryptophan, the amino acid precursor of serotonin. Secondary goals are to determine how this experimental manipulation influences people's feelings as well as their perceptions of other's social behaviour following interpersonal events, and social cognitions at the end of the day. An exploratory goal is to investigate if these effects are moderated by genes thought to be involved in MDD.

The primary hypothesis to be tested is that tryptophan will reduce quarrelsome behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* At least one first-degree family member with MDD
* Willingness to cooperate; to sign written informed consent

Exclusion Criteria:

* Any current or past MDD or other mood disorder as determined by the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID)
* Any current anxiety disorder, psychotic disorder, substance use disorder, eating disorder, or somatoform disorder as determined by SCID
* Any contraindication for the use of tryptophan, i.e. pregnancy, diabetes, cancer or a history of cancer, a history of any scleroderma-like condition, evidence of achlorhydria, upper bowel malabsorption, or irritation of the urinary bladder
* Current use of psychotropic medications including medications for psychiatric problems (e.g., antidepressants such as Mono Amine Oxidase inhibitors and fluoxetine) or migraines
* Not speaking Dutch fluently

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
quarrelsome behaviour | 28 days
  quarrelsome behaviour is measured daily for 28 days using Ecological Momentary Assessment.

SECONDARY OUTCOMES:
interpersonal behaviour | 28 days
  measures are assessed on a daily basis for 28 days with ecological momentary assessment
affect | 28 days
  measures are assessed on a daily basis for 28 days with ecological momentary assessment
perceptions of others | 28 days
  measures are assessed on a daily basis for 28 days with ecological momentary assessment
social cognitions | 28 days
  measures are assessed daily for 28 days with ecological momentary assessment

OTHER OUTCOMES:
Serotonin transporter polymorphism | 1 day
  Prior to starting the 28 days of social interacton recording participants are instructed about the study procedures. The saliva samples are analyzed for Serotonin transporter polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Marije aan het Rot, Dr., Principal Investigator — University of Groningen